CLINICAL TRIAL: NCT00886626
Title: GLP-1 Therapy for Weight Loss and Improved Glucose Tolerance in Obese Children: A Randomized, Controlled, Pilot Study
Brief Title: GLP-1 Therapy for Weight Loss and Improved Glucose Tolerance in Obese Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0902M59181
Record Dates: First submitted 2009-04-22; First posted 2009-04-23 (Estimated); Results first posted 2012-08-17 (Estimated); Last update posted 2012-10-29 (Estimated); Status verified 2012-10

CONDITIONS: Obesity, Morbid
Keywords: Obesity; Impaired Glucose Tolerance; Children
MeSH Terms: conditions — Obesity, Morbid; Obesity; Glucose Intolerance | interventions — Exenatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exenatide (Experimental): Exenatide
  Interventions: Drug: Exenatide
- Control (No Intervention): Control - no intervention

INTERVENTIONS:
Drug: Exenatide — Exenatide, subcutaneous injection, 10 mcg, twice per day
  Other Names: Byetta
  Arms: Exenatide

SUMMARY:
The prevalence of severely obese children is on the rise. Behavioral therapies for weight loss are successful in some, but others need more aggressive approaches such as drug therapy. In addition, up to 25% of severely obese children have impaired glucose tolerance (IGT), which places them at significantly elevated risk of developing type 2 diabetes mellitus and cardiovascular disease. Although various drug therapies for weight loss and IGT have been explored in adults, few have been evaluated in children.

Recently, a new drug class has emerged that targets deficiencies of GLP-1. One of the main glycemic mechanisms of action of the GLP-1 agonists such as exenatide is to enhance glucose disposal in the postprandial setting and improve glucose tolerance. In addition, exenatide can induce weight loss by decreasing appetite and slowing gastric motility.

DETAILED DESCRIPTION:
This will be a randomized, open-label, controlled, crossover clinical trial in 12 patients. All patients will receive exenatide and undergo the control phase. Following baseline testing, participants will be randomly assigned to treatment order: therapy (exenatide) or control (lifestyle modification). Half (n = 6) will receive exenatide first (3-months) then cross over to control (no drug therapy for 3-months). Half (n = 6) will be assigned to control first (3-months) then cross over to exenatide (3-months). All efforts will be made to stratify randomization based on gender of the participants. Treatment and control conditions will be three months each. Because of the route of administration of exenatide (subcutaneous injection), placebo will not be utilized for the control phase of the study.

Participants in this study will engage in background intensive lifestyle modification offered by the University of Minnesota Pediatric Weight Management Clinic for the entire study, even during the active drug treatment phase. Intensive lifestyle modification will be purely clinical in nature in which children and their families receive continuing counseling from a team of trained professionals including physicians, dieticians, and psychologists to reduce weight by making healthier eating choices and increasing physical activity.

The screening visit will take place in the Pediatric Weight Management Clinic and will include a complete medical history and physical examination. Screening will include review of medical records for previous clinical and laboratory data (including clinically-ordered glucose tolerance test results). All research testing will take place in the University of Minnesota General Clinical Research Center (GCRC). Subjects will undergo testing at the following intervals: baseline, immediately after the first 3-month phase (whether exenatide or control), and immediately after the second 3- month phase (whether exenatide or control). The following measures will be collected after the subject has been fasting for at least twelve hours:

* Height, weight, body mass index, waist and hip circumference
* Fat and lean mass (dual energy x-ray absorptiometry: DXA)
* Tanner stage determination (performed during screening physical exam or may be obtained from medical chart)
* Fasting lipid profile (total-, LDL-, and HDL-cholesterol, triglycerides)
* Systolic and diastolic blood pressure
* Oral glucose tolerance test (glucose and insulin measured every 30 minutes for 2 hours)
* Endothelial function (digital reactive hyperemia: EndoPAT 2000, Itamar Medical) - in addition to the baseline measure, endothelial function testing will occur at hours one and two of the oral glucose tolerance test
* Frozen plasma for storage - in addition to the baseline blood draw, blood for endothelial biomarkers will be obtained at hours one and two of the oral glucose tolerance test
* Arterial stiffness (pulse wave velocity; augmentation index: Sphygmocor, AtCor Medical)
* Frozen plasma for pharmacokinetic determination of exenatide in children

ELIGIBILITY:
Inclusion Criteria:

* Age 8-19 years old
* Subject able to give assent, and parent/guardian capable of giving consent on behalf of the child
* Body mass index (BMI) ≥ 99th percentile (based on gender and age)

Exclusion Criteria:

* Type 1 or 2 diabetes mellitus
* Initiation of a new drug therapy within the past 30 days prior to the screening visit
* BMI ≥ 55
* History of weight loss surgery
* Obesity from a genetic cause (e.g., Prader-Willi)
* Central nervous system injury or severe neurological impairment
* Known systolic or diastolic dysfunction or heart failure
* Females who are currently pregnant or planning to become pregnant
* Liver enzymes > 2.5 times upper limit of normal
* Severe renal impairment (defined as creatinine clearance <30 mL/min)
* Gastrointestinal disease

Ages: 8 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2009-05; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron S. Kelly, Ph.D., Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Kelly AS, Metzig AM, Rudser KD, Fitch AK, Fox CK, Nathan BM, Deering MM, Schwartz BL, Abuzzahab MJ, Gandrud LM, Moran A, Billington CJ, Schwarzenberg SJ. Exenatide as a weight-loss therapy in extreme pediatric obesity: a randomized, controlled pilot study. Obesity (Silver Spring). 2012 Feb;20(2):364-70. doi: 10.1038/oby.2011.337. Epub 2011 Nov 10. PMID 22076596

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred from October 2009 - August 2010; participants were recruited from medical clinics in the Minneapolis-St. Paul area.
Pre-assignment Details: 29 patients qualified for the study and were approached about participation. 12 agreed to participate.
Groups:
- Exenatide Then Control: Exenatide 5 mcg for 1-month then uptitration to 10-mcg for remaining 2-months followed by control for 3-months
- Control Then Exenatide: No medication control for 3-months then exenatide 5 mcg for 1-month uptitrated to 10 mcg for following 2-months
Period: Period 1 (90 Days)
Arm/Group | Exenatide Then Control | Control Then Exenatide
Started | 6 | 6
Completed | 5 | 6
Not Completed | 1 | 0
Period: Period 2 (90 Days)
Arm/Group | Exenatide Then Control | Control Then Exenatide
Started | 5 | 6
Completed | 5 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All enrolled participants
Arm/Group | All Participants
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12
  Between 18 and 65 years | 0
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 12.7 (2.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Mass Index (BMI)
Description: Change in body mass index (BMI) over three months
Time Frame: 3-month
Population: Data from all participants who completed the trial were analyzed.
Measure: Mean (Standard Deviation); unit: change in kg/m^2
Groups:
- Exenatide: Exenatide 5 mcg for 1-month then up-titration to 10-mcg for remaining 2-months. Participants came from period 1 and period 2.
- Control: No medication control for 3-months. Participants came from period 1 and period 2.
Arm/Group | Exenatide | Control
Number analyzed (Participants) | 11 | 11
change in kg/m^2 | -0.9 (1.2) | 0.84 (1.3)

ADVERSE EVENTS:
Time Frame: 6-month
Description: Adverse Events were evaluated over length of study (6 months; 180 days)
Groups:
- Exenatide: Exenatide 5 mcg for 1-month then uptitration to 10-mcg for remaining 2-months.
- Control: No medication control for 3-months.
Arm/Group | Exenatide | Control
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 4/11 | 0/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exenatide (N=11) | Control (N=11)
Nausea (Gastrointestinal disorders) | 4 (4) | 0 (0)

LIMITATIONS AND CAVEATS:
Small sample size; un-blinded; crossover study design

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No